CLINICAL TRIAL: NCT04562506
Title: Repetitive Transcranial Magnetic Stimulation With H-coil in Alzheimer's Disease: A Double-blind, Placebo-controlled Pilot Study
Brief Title: Repetitive Transcranial Magnetic Stimulation With H-coil in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giancarlo Comi (Other)
Responsible Party: Sponsor-Investigator, Giancarlo Comi, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMS-AD
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS stimulation (Active Comparator): real deep excitatory, high frequency rTMS with H-coil stimulation
  Interventions: Device: rTMS with H-coil
- Sham rTMS stimulation (Sham Comparator): sham high frequency H-coil stimulation
  Interventions: Device: Sham rTMS stimulation with H-coil

INTERVENTIONS:
Device: rTMS with H-coil — Deep repetitive transcranial manetic stimulation or sham stimulation with H-coil
  Arms: Real rTMS stimulation
Device: Sham rTMS stimulation with H-coil — Sham rTMS stimulation
  Arms: Sham rTMS stimulation

SUMMARY:
Focal repetitive transcranial magnetic stimulation (rTMS) has been applied to improve cognition in Alzheimer's disease (AD) with conflicting results. In this study we aimed to explore feasibility, safety and efficacy of excitatory rTMS of bilateral DLPFC applied with H-coil in AD in a pilot randomized, placebo-controlled, double-blind study.

DETAILED DESCRIPTION:
Study Design The study was a double-blind, placebo-controlled paradigm, with randomization into a real rTMS group or a sham rTMS

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risk of the study and provide signed and dated informed consent.
* Male or female subjects, 18 to 80 years old.
* Diagnosis of Alzheimer's disease according to the DSM IV
* Subjects who answered all questions in the TMS pre-treatment safety questionnaire in a negative manner.
* Have given written informed consent

Exclusion Criteria:

* Presence of an additional neurological or psychiatric pathology.
* Severe personality disorder.
* Uncontrolled hypertension.
* History of epilepsy, seizures, febrile convulsions.
* History of epilepsy or seizures in first degree relatives.
* History of head injury or stroke.
* Presence of metal prostheses in the head (except dental fillings).
* Metal implants or known history of any metal particles in the eye, cardiac pacemakers, cochlear implants, use of neurostimulators or medical pumps.
* History of migraine within the past six months.
* History of drug or alcohol abuse.
* Impossibility of adequate communication with the examiner.
* Participation in another clinical study, either concomitant or within the previous 3 months.
* Inability to sign the consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-09-08 (Actual)

PRIMARY OUTCOMES:
Improvement at Alzheimer's Disease Assessment Scale-cognitive over time | Change in the score between Baseline evaluation and end of the treatment (2 months after start of the treatment)
  Brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia

SECONDARY OUTCOMES:
Improvement at Mini Mental State Examination scale over time | Baseline evaluation, 1 month after start of the treatment, end of the treatment (2 months after start of the treatment) and end of follow-up (4 months after start of the treatment)
  Neuropsychological test used to assess the intellectual efficiency disorders and the presence of cognitive impairment
Improvement at Beck Depression Inventory scale-II over time | Baseline evaluation, 1 month after start of the treatment, end of the treatment (2 months after start of the treatment) and end of follow-up (4 months after start of the treatment)
  Self-report inventory, psychometric test used to assess the severity of depression
Improvement at Clinical Global Impression-Improvement scale over time | Baseline evaluation, 1 month after start of the treatment, end of the treatment (2 months after start of the treatment) and end of follow-up (4 months after start of the treatment)
  Scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention
Persistence of improvement at Alzheimer's Disease Assessment Scale-cognitive over time | Change in the score between end of treatment (2 months after start of the treatment) and end of follow-up (4 months after start of treatment)
  Brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: ICF, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: data are available from the corresponding author, upon reasonable request.

REFERENCES:
- [Derived] Leocani L, Dalla Costa G, Coppi E, Santangelo R, Pisa M, Ferrari L, Bernasconi MP, Falautano M, Zangen A, Magnani G, Comi G. Repetitive Transcranial Magnetic Stimulation With H-Coil in Alzheimer's Disease: A Double-Blind, Placebo-Controlled Pilot Study. Front Neurol. 2021 Feb 18;11:614351. doi: 10.3389/fneur.2020.614351. eCollection 2020. PMID 33679572